CLINICAL TRIAL: NCT03369132
Title: Efficacy of Natural Seawater Based Throat Spray in Acute Sore Throat Relief: a Prospective, Randomized, Double-blind, Placebo-controlled, Multicentre Clinical Study
Brief Title: Efficacy of Natural Seawater Based Throat Spray in Acute Sore Throat Relief
Acronym: FLASH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laboratoire de la Mer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FLASH-CZ-2017-01
Record Dates: First submitted 2017-11-16; First posted 2017-12-11 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Sore Throat
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Angiflash (Experimental)
  Interventions: Device: Angiflash
- Placebo (Placebo Comparator)
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Angiflash — throat spray (20 ml) containing hypertonic seawater, vegetable glycerin, natural mint, acacia honey, propolis extract, essential oils of thyme linalool, ravintsara and wintergreen, natural lemon flavor.
  Other Names: Seawater based throat spray
  Arms: Angiflash
Device: Placebo — water based throat spray matching Angiflash for posology, dispensed volume, shape and size.
  Other Names: Placebo throat spray
  Arms: Placebo

SUMMARY:
Prospective, randomized, double-blind, placebo-controlled, multicentre clinical trial to assess the efficacy and tolerability of natural seawater based throat spray among adult patients with acute sore throat.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adults (male or female) aged ≥ 18 years old.
* 2. Patients with complaint of sore throat ≤ 72h.
* 3. Sore throat exclusively due to upper respiratory tract infection (tonsillitis, pharyngitis, rhinopharyngitis).
* 4. Clinical confirmation by the physician for the presence of typical signs (spontaneous pain, local inflammation) of acute pharyngitis or tonsillitis.
* 5. Pain intensity scored by patient on the 5-point descriptive pain intensity scale as slight, mild or moderate.
* 6. Willingness to provide written informed consent prior to perform of any study related procedure.
* 7. Subjects agreeing to follow the study requirements during the whole study period (including forbidden medication and food supplements).
* 8. Subjects agreeing not to modify their lifestyle habits during the whole study period (diet, physical activity).
* 9. Subject affiliated to social security.
* 10. Subject able to understand verbal and written local language and in capacity to fill-in patient diary by himself/herself.

Exclusion Criteria:

* 1. Previous history of allergy or known intolerance to one of the following formulation ingredients: seawater, vegetable glycerin, mint, lemon, acacia honey, propolis, essential oils.
* 2. Active Smokers.
* 3. Fever > 38°C at randomization.
* 4. Past or current throat phlegmon.
* 5. Past or current seasonal allergy.
* 6. Past or current asthma.
* 7. Past or current chronic rhinosinusitis.
* 8. Past or current chronic obstructive pulmonary disease (COPD).
* 9. Past or current ENT (Ear, Nose and Throat) cancer.
* 10. Acute rhinosinusitis.
* 11. Controlled or uncontrolled diabetes.
* 12. Gastroesophageal reflux disease (GERD).
* 13. Known immunodeficiency.
* 14. Any painful condition that may distract attention from sore throat pain (ex: mouth ulcers etc.) or that requires analgesic usage.
* 15. Any disease that may interfere with the study aim from investigator's opinion.
* 16. Evidence of mouth breathing or severe coughing.
* 17. Patient with severe pain intensity on 5-point descriptive pain intensity scale.
* 18. Subjects taking:

  * chronic treatment for throat or other ENT pathology,
  * current antibiotherapy or stopped less than 2 weeks before inclusion,
  * chronic treatment (>3 months) with local or systemic corticotherapy, or immunotherapy,
  * local or systemic antihistaminic.
* 19. Subjects refusing to stop at entry into the study:

  * throat spray, lozenge, pastille,
  * local throat or systemic analgesic,
  * medicated confectionary,
  * nasal wash and spray,
  * nasal corticosteroid or antihistaminic nasal spray,
  * medication to gargle,
  * honey, propolis, or any sore throat home remedies.
* 20. Known liver disease or hypersensitivity to paracetamol.
* 21. Pregnant, breastfeeding or seeking pregnancy women.
* 22. Positive result from rapid strep throat test.
* 23. Subjects already included once in this study.
* 24. Subjects participating in another clinical trial or in the exclusion period to another study.
* 25. Subjects having a member of his/her home who is currently participating to this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2017-11-06 (Actual); Primary Completion 2018-05-31 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Sore Throat Relief | Over the first three days
  Evaluation of sore throat relief using the 7-point sore throat relief scale (STRS)

SECONDARY OUTCOMES:
Sore Throat Individual Symptoms Relief | Day 1, 2, 3, 4, 5, 5, 7 to 8.
  Evaluation of relief of sore throat individual symptoms (dry throat, burning/painful sensation, hoarseness/husky voice, painful talk, painful swallowing, irritation, prickly sensation/tingle, scratchy/itchy throat) using a 10-point rating scale
Sore Throat Pain Intensity | Day 1, 2, 3, 4, 5, 5, 7 to 8.
  Change from baseline of the Sore Throat Pain Intensity using a Visual Analog Scale (VAS) (STPIS)
Difficulty Swallowing | Day 1, 2, 3, 4, 5, 5, 7 to 8.
  Change from baseline of the difficulty of swallowing using a VAS (DSS)
Swollen Throat | Day 1, 2, 3, 4, 5, 5, 7 to 8.
  Change from baseline of the swollen throat using a VAS (SwoTS)
Overall efficacy assessed by the physician | Day 8
  Overall efficacy assessed by the physician using a 5-point descriptive scale
Compliance: assessment of the number of use per day and the number of spray per use | Day 1, 2, 3, 4, 5, 5, 7 to 8.
  Assessment of the patient usage: frequency per day and number of spray per use
Product Satisfaction | Day 8
  Assessment of the overall satisfaction using a 5-point descriptive scale
Incidence of adverse events occuring during the study | Day 1, 2, 3, 4, 5, 5, 7 to 8.
  Number of adverse events and serious events occuring during the study and evaluation of the severity and causality.

CONTACTS AND LOCATIONS:
Overall Officials: Ivana Skardova, M.D., Principal Investigator — MEDIGATE care s.r.o
Locations (16):
- Czechia (16):
  - MUDr. Lenka Dybova, Brno
  - MUDr. Libor Hemzsky, Choltice
  - NEFROMED s.r.o., Dejvice
  - MEDIGATE care s.r.o, Hradec Králové
  - MUDr. Petra Hoskova, Hradec Králové
  - MUDr. Jana Dvorakova s.r.o., Hradec Králové
  - MUDr. Danuse Mikeschova, Karlovy Vary
  - Azita s.r.o., Malšice
  - Fortmedica s.r.o., Prague
  - GM ordinace s.r.o, Prague
  - MUDr Sylva Kohoutova, Prague
  - Ordinace Optima s.r.o, Prague
  - MUDr. Lenka Fejfarova, Prague
  - Saniga s.r.o., Sokolov
  - MUDr. Jan Bartusek, Teplice
  - A-MEDICOS s.r.o., Zlín

IPD SHARING:
Plan to Share IPD: No